CLINICAL TRIAL: NCT01891604
Title: Study the Safety and Efficacy of Probiotics Use in Premature Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Never Initiated due to Impact approval from institution not being obtinaed
Sponsor: University of Manitoba (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Principal Investigator, Dr. James Friel, Professor, University of Manitoba
Model: Parallel
Other Study IDs: jamesfriel2013
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases | interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: breast milk with Bifidobacterium Longum subp. Infantis R0033
Dietary Supplement: breast milk

SUMMARY:
Prophylactic enteral probiotics may enhance clinical markers and biomarkers of preterm infants' health, and may also play a role in reducing NEC and associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* born with weight<1500 g
* hospitalized within 48 hours after birth

Exclusion Criteria:

* present with evidence or suspicion of congenital intestinal obstruction
* perforation
* gastroschisis
* large omphalocele
* congenital diaphragmatic hernia
* major congenital heart defects

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Calprotectin will be used to determine the effect for probiotics | day1 and day30 of the observation